CLINICAL TRIAL: NCT05020769
Title: A Phase II/III Clinical Study to Evaluate the Efficacy and Safety of SI-B001 in Combination With Osimertinib Mesylate Tablets in the Treatment of Recurrent and Metastatic Non- Small Cell Lung Cancer
Brief Title: SI-B001 Combined With Osimertinib Mesylate Tablets in the Treatment of Recurrent Metastatic Non-small Cell Lung Cancer.
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001_210
Record Dates: First submitted 2021-08-22; First posted 2021-08-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SI-B001 combined with osimertinib_A (Experimental): Patients with locally advanced/metastatic NSCLC progressed on 3rd generation EGFR-TKI treatment.
  Interventions: Drug: SI-B001; Drug: Osimertinib
- SI-B001 combined with osimertinib_B (Experimental): Patients with locally advanced/metastatic NSCLC progressed on prior EGFR-TKI treatment and with T790M negative mutation.
  Interventions: Drug: SI-B001; Drug: Osimertinib
- SI-B001 combined with osimertinib_C (Experimental): Patients with locally advanced/metastatic NSCLC and with EGFR exon20ins mutation.
  Interventions: Drug: SI-B001; Drug: Osimertinib

INTERVENTIONS:
Drug: SI-B001 — SI-B001 is administered by intravenous drip once weekly (QW). 120 min ± 10 min after the first intravenous drip, if the infusion reaction is tolerable during the first dose, the subsequent infusion can be completed within 60-120 min (unless agreed or required by the investigator, the infusion time can be extended).
Drug: Osimertinib — Osimertinib is administered at the recommended dose of 80mg daily.

SUMMARY:
This multi-center, open label Phase II/III clinical study is performed in patients with locally advanced/metastatic NSCLC progressed on prior EGFR-TKI treatment or with non TKI-sensitizing mutation or patients with EGFR exon20ins mutation. This study is investigating the safety and efficacy of SI-B001 at monotherapy RP2D or lower combined with Osimertinib in patients with locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Male or female;
3. Age: ≥ 18 years;
4. Expected survival time ≥ 3 months;
5. Patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) confirmed by histopathology and/or cytology, T790M-negative, Exon20ins mutation resistant to the third generation EGFR TKI after the first or second line treatment, or resistance to the first or second generation TKI after the first line treatment;
6. Consent to provide an archived tumor tissue specimen or fresh tissue sample (an FFPE block or approximately 6-12 white slides with a size of 5μm) from the primary or metastatic tumor within 6 months of the date of consent. Participants who were unable to provide tumor tissue samples could be enrolled if they met other inclusion and exclusion criteria after evaluation by investigators.
7. Must have at least one measurable lesion as defined by RECISTv1.1;
8. Performance status score ECOG0 or 1;
9. Toxicity from previous antineochemical therapy has returned to grade 1 or less as defined by NCI-CTCAE v5.0 (asymptomatic laboratory abnormalities such as elevated ALP, hyperuricemia, elevated serum amylase/lipase, and elevated blood glucose were considered by the investigator, and toxicity with no safety risk was judged by the investigator; Except for alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stable with hormone replacement therapy).
10. No severe cardiac dysfunction, left ventricular score ≥ 50%;
11. The level of organ function must meet the following criteria:

    1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count ≥ 80 × 10^9/L, hemoglobin ≥ 90 g/L;
    2. Liver function: TBIL ≤ 1.5ULN (total bilirubin ≤ 3ULN for subjects with Gilbert's syndrome, liver cancer or liver metastases); AST and ALT ≤ 2.5ULN for subjects without liver metastases; AST and ALT ≤ 5.0ULN for subjects with liver metastases;
    3. Renal function: creatinine (Cr) ≤ 1.5ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (according to CockcroftandGault formula).
12. Coagulation function: international normalized ratio (INR) ≤ 1.5 × ULN, and activated partial thromboplastin time (APTT) ≤ 1.5ULN;
13. Urine protein ≤ 2 + (measured by dipstick) or < 1000 mg/24 h (urine);
14. Premenopausal women of childbearing potential must have a negative serum or urine pregnancy test 7 before starting treatment and must be non-lactating; all patients (male or female) should take adequate barrier contraception measures throughout the treatment cycle and 6 months after the end of treatment.

Exclusion Criteria:

1. Gene sequencing showed that there were MET, ALK, RET, HER2 and other driver gene mutations related to the occurrence and development of tumors.
2. Patients with prior systemic chemotherapy as part of first - or second-line systemic therapy;
3. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, and major surgery were used within 4 weeks before the first dose, and palliative radiotherapy, targeted therapy (including small molecule tyrosine kinase inhibitors), and other anti-tumor treatments were used within 2 weeks before the first dose.
4. The history of severe heart disease within the past six months was screened, such as symptomatic congestive heart failure (CHF) ≥ grade 2 (CTCAE v5.0), New York Heart Association (NYHA) ≥ grade 2 heart failure, acute coronary syndrome, etc.
5. Prolonged QT interval (QTc > 450 msec in men or QTc > 470 msec in women), complete left bundle branch block, atrioventricular block III degree;
6. Active autoimmune and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory intestinal diseases and Hashimoto's thyroiditis, etc., excluding type I diabetes mellitus, hypothyroidism that can be controlled only by replacement therapy, and skin diseases without systemic treatment (such as vitiligo and psoriasis);
7. Other malignant tumors diagnosed within 5 years before the first dose of treatment, except those with radical basal cell carcinoma, squamous cell carcinoma of the skin, and/or radical resection in situ carcinoma considered by investigators to be eligible;
8. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg);
9. Pulmonary disease grade ≥3 was defined according to CTCAE v5.0, including dyspnea at rest, or requiring continuous oxygen therapy, or a history of interstitial lung disease (ILD).
10. There were symptoms of active central nervous system metastasis. However, patients with stable parenchymal metastases could be enrolled, and whether they were stable was defined by the investigators.
11. Patients with a history of allergy to the recombinant humanized or human-mouse chimeric antibody or to SI-B001 or any of the excipients of the chemotherapeutic agents used in this trial;
12. A history of autologous or allogeneic stem cell transplantation;
13. The cumulative dose of anthracyclines in previous (new) adjuvant therapy was > 360 mg/m^2;
14. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 10^4) or hepatitis C virus infection (HCV-RNA > the lower limit of detection in the research center);
15. Active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc.;
16. Received other unmarketed investigational drugs or treatments within 4 weeks before study enrollment;
17. Other conditions for trial participation were not considered by the investigator to be appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 24 months
  Objective Response Rate
Optimal combination dose (only Phase IIa) | Up to approximately 24 months
  Optimal combination dose for SI-B001 and Osimertinib (only IIa)

SECONDARY OUTCOMES:
PFS | Up to approximately 24 months
  Progression-free Survival
DCR | Up to approximately 24 months
  Disease Control Rate
DOR | Up to approximately 24 months
  Duration of Response
TEAE | Up to approximately 24 months
  Treatment Emergent Adverse Events
Cmax | Up to approximately 24 months
  Maximum serum concentration
Tmax | Up to approximately 24 months
  Time to maximum serum concentration
Ctrough | Up to approximately 24 months
  Minimum serum concentration
ADA | Up to approximately 24 months
  anti-SI-B001 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University Cancer Center (SYSUCC)
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangdong, Guangzhou